CLINICAL TRIAL: NCT02347878
Title: Self-control Trial to Evaluate the Role of Aprepitant in the Prophylaxis of Post-lumbar-punture-headache (PLPH)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Liang Wang, Doctor, Sun Yat-sen University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PLPH
Record Dates: First submitted 2015-01-21; First posted 2015-01-27 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Leukemia; Lymphoma
Keywords: leukemia; lymphoma; lumbar puncture; intrathecal treatment; post-lumbar puncture headache
MeSH Terms: conditions — Leukemia; Lymphoma; Post-Dural Puncture Headache | interventions — Aprepitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment arm (Experimental): this treatment arm will received aprepitant 1 hour before lumbar puncture and intrathecal treatment.
  Interventions: Drug: Aprepitant
- control arm (No Intervention): this arm will received nothing 1 hour before lumbar puncture

INTERVENTIONS:
Drug: Aprepitant — use aprepitant 1 hour before lumbar puncture and intrathecal treatment
  Other Names: Emend
  Arms: treatment arm

SUMMARY:
Headache following a lumbar puncture （post-lumbar-puncture headache,PLPH）is a common and often debilitating syndrome, which was reported to occur in about 40% patients who received lumbar puncture. Now there lacks of effective approaches in the prophylaxis of PLPH, although some physicians consider bed rest for at least 6 hours to be a useful methods (Some recent meta-analysis found no benefit of bed rest for any hours in the prevention of PLPH). Studies have found that P substances and its receptor (Neurokinin-1 receptor, NK-1R)have played an important role in the pathogenesis of PLPH. Thus, we hypothesize that use of NK-1R inhibitor (aprepitant) 1 hour before lumbar puncture may decrease the incidence of PLPH and lower the severity of PLPH.

DETAILED DESCRIPTION:
Headache following a lumbar puncture （post-lumbar-puncture headache,PLPH）is a common and often debilitating syndrome, which was reported to occur in about 40% patients who received lumbar puncture. Now there lacks of effective approaches in the prophylaxis of PLPH, although some physicians consider bed rest for at least 6 hours to be a useful methods (Some recent meta-analysis found no benefit of bed rest for any hours in the prevention of PLPH). Studies have found that P substances and its receptor (Neurokinin-1 receptor, NK-1R)have played an important role in the pathogenesis of PLPH. Thus, we hypothesize that use of NK-1R inhibitor (aprepitant) 1 hour before lumbar puncture may decrease the incidence of PLPH and lower the severity of PLPH.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as acute leukemia, or lymphoma
* Patients will received repeated lumbar puncture (at least 2 times, and at least 2 weeks apart) and intrathecal treatment
* Without CNS involvement
* Without headache for at least 1 week before the day of lumbar puncture
* The platelet count was at least 30×10e9/L

Exclusion Criteria:

* With CNS involvement of disease
* With headache before lumbar puncture
* Needs lumbar puncture more than once a week

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
incidence of any grade post-lumbar-puncture headache | date from the day of lumbar puncture to 2 weeks after lumbar puncture

SECONDARY OUTCOMES:
incidence of grade 3/4 post-lumbar-puncture headache | date from the day of lumbar puncture to 2 weeks after lumbar puncture

CONTACTS AND LOCATIONS:
Overall Officials: Liang Wang, DOCTOR, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China